CLINICAL TRIAL: NCT06866808
Title: Combined Effects of Talocrural Mobilization With Movement and Therapeutic Ultrasound on Pain, Balance and Disability in Athletes With Ankle Sprain.
Brief Title: Combined Effects of Talocrural MWM and Therapeutic US on Pain, Balance and Disability in Athletes With Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aman Naveed
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group receive Talocrural mobilization with therapeutic ultrasound therapy.
  Interventions: Other: talocrural MWM and Therapeutic US
- Control Group (Other): Control Group receive the conventional physiotherapy treatment including icing and ankle isometrics.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: talocrural MWM and Therapeutic US — Mobilization with movement alongwith the therapeutic ultrasound
  Arms: Experimental Group
Other: Conventional physiotherapy — Ankle isometrics, calf stretches, icing
  Arms: Control Group

SUMMARY:
Combined Effects of Talocrural MWM and Therapeutic US on Pain, Balance and Disability in Athletes With Ankle Sprain. Study consist of two groups. One group receives conventional physiotherapy treatment conventional physiotherapy treatment including icing and ankle isometrics. Other receives Talocrural mobilization with therapeutic ultrasound therapy on ankle joint.

DETAILED DESCRIPTION:
Ankle sprain is a prevalent injury marked by harm to the ligaments that provide support to the ankle joint. Ligaments are resilient and pliable fibrous structures that establish a connection between bones, providing joint stability. Ankle sprains commonly arise from excessive rotation or bending of the foot, resulting in the stretching or tearing of ligaments. Talocrural mobilization is a therapy method that utilizes manual techniques to treat the Talocrural joint, which is the joint formed by the tibia, fibula, and talus bone in the ankle. This mobilization approach is designed to enhance joint function, expand range of motion, and alleviate symptoms related to limited movement or musculoskeletal disorders that impact the ankle joint.

Randomized Control Trial will be conducted at the Punjab Stadium over a 10-month period. The sample size, after considering a 10% attrition rate, will consist of 15 participants in each group. Group A, the control group, will receive conventional physiotherapy treatment including icing and ankle isometrics, while Group B will undergo Talocrural mobilization with therapeutic ultrasound therapy and conventional physiotherapy. Participants aged 18 to 40 years diagnosed with ankle sprain and experiencing ankle pain within the last six weeks will be included. Exclusion criteria involve a history of ankle or foot fractures, concurrent lower extremity injuries, neurological disorders affecting lower limb function, and recent ankle or foot surgeries within the last six months. Data collection tools include the Foot and Ankle Disability Index (FADI) for disability, Star Excursion Balance Test (SEBT) for balance, and Numeric Pain Rating Scale (NPRS) for pain intensity. The study will involve pre and post assessments over a 6-week duration, analyzing changes within and between groups using statistical tests such as paired sample t-test, Wilcoxon signed rank test, independent sample t-test, and Mann Whitney U test. The Talocrural mobilization protocol for Group B will comprise five sessions per week, each lasting 40 minutes, including 20 minutes of therapeutic ultrasound and 20 minutes of Talocrural mobilization. The data will be analyzed using SSP for Windows software version 25.

ELIGIBILITY:
Inclusion Criteria:

* Athletes age 18 to 40 years
* Patients diagnosed with ankle sprain.
* Onset of ankle pain during last six weeks.

Exclusion Criteria:

* Previous history of ankle or foot fractures.
* Concurrent lower extremity injuries affecting pain, balance, and disability assessment
* Any neurological disorders affecting lower limb function.
* Recent ankle or foot surgeries within the last six months.
* Planned surgeries in next 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Athlete disability index | 6 weeks
  The Athlete Disability Index (ADI) is a self-administered questionnaire specifically designed to assess the level of disability experienced by athletes due to low back pain (LBP)
Berg balance scale | 6 weeks
  The Berg Balance Scale (BBS) is a popular clinical tool for assessing balance and fall risk in older persons. Katherine Berg created it to assess balance during various activities.
Numeric Pain Rating Scale (NPRS) | 6 weeks
  The Numeric Pain Rating Scale (NPRS) is a widely used tool for assessing subjective experiences, particularly pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, MS, Principal Investigator — Riphah International University
Locations (1):
- Punjab Stadium, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ersoy U, Kocak UZ, Unuvar E, Unver B. The Acute Effect of Talocrural Joint Mobilization on Dorsiflexor Muscle Strength in Healthy Individuals: A Randomized Controlled Single-Blind Study. J Sport Rehabil. 2019 Aug 1;28(6):601-605. doi: 10.1123/jsr.2018-0124. PMID 30040011
- [Background] Kaminski TW, Needle AR, Delahunt E. Prevention of Lateral Ankle Sprains. J Athl Train. 2019 Jun;54(6):650-661. doi: 10.4085/1062-6050-487-17. Epub 2019 May 22. PMID 31116041
- [Background] D'Hooghe P, Cruz F, Alkhelaifi K. Return to Play After a Lateral Ligament Ankle Sprain. Curr Rev Musculoskelet Med. 2020 Jun;13(3):281-288. doi: 10.1007/s12178-020-09631-1. PMID 32377961
- [Background] Chen ET, Borg-Stein J, McInnis KC. Ankle Sprains: Evaluation, Rehabilitation, and Prevention. Curr Sports Med Rep. 2019 Jun;18(6):217-223. doi: 10.1249/JSR.0000000000000603. PMID 31385837
- [Background] Sarcon AK, Heyrani N, Giza E, Kreulen C. Lateral Ankle Sprain and Chronic Ankle Instability. Foot Ankle Orthop. 2019 Jun 13;4(2):2473011419846938. doi: 10.1177/2473011419846938. eCollection 2019 Apr. PMID 35097325
- [Background] Medina McKeon JM, Hoch MC. The Ankle-Joint Complex: A Kinesiologic Approach to Lateral Ankle Sprains. J Athl Train. 2019 Jun;54(6):589-602. doi: 10.4085/1062-6050-472-17. Epub 2019 Jun 11. PMID 31184957
- [Background] Halabchi F, Hassabi M. Acute ankle sprain in athletes: Clinical aspects and algorithmic approach. World J Orthop. 2020 Dec 18;11(12):534-558. doi: 10.5312/wjo.v11.i12.534. eCollection 2020 Dec 18. PMID 33362991
- [Background] Herzog MM, Kerr ZY, Marshall SW, Wikstrom EA. Epidemiology of Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):603-610. doi: 10.4085/1062-6050-447-17. Epub 2019 May 28. PMID 31135209